CLINICAL TRIAL: NCT06752304
Title: A Longitudinal Study of Severe and Enduring Eating Disorders
Acronym: Long-SEED
Status: Recruiting | Type: Observational
Sponsor: Uppsala University Hospital (Other)
Collaborators: Forte (Industry); The Söderström König Foundation (Unknown); Fonden för psykisk hälsa (Unknown)
Responsible Party: Principal Investigator, Martina Isaksson, PhD, clinical researcher, Uppsala University Hospital
Other Study IDs: Long-SEED
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge Eating Disorder; Other Specified Feeding or Eating Disorder
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Blood samples for analyses of hormones and inflammatory markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adolescent ED cohort
- Adult ED cohort

SUMMARY:
The goal of this observational longitudinal study is to investigate characteristics and factors associated with the development of Severe and Enduring Eating Disorders (SEED). In this project, the researchers will follow two prospective cohorts of patients with eating disorders (ED), one adolescent (ages 14-17) and one adult (ages 18+), in terms of change in and impact of clinical, psychological, and biological risk factors.

Data will be collected at baseline, after treatment, two years after baseline, and thereafter five, 10 and 20 years after baseline. Participants will be asked to undergo a physical examination, leave blood samples, be interviewed, and fill in questionnaires. If the participants are minors, their care takers will also fill in the questionnaires.

The study aims to explore how clinical, psychological, and biological risk factors-including comorbidity, personality characteristics, difficulties with emotion regulation (ER), cognitive inflexibility, loneliness, severe ED symptoms, and inflammatory activation-contribute to a chronic course of the disorder.

DETAILED DESCRIPTION:
BACKGROUND, AIMS AND HYPOTHESES

Eating disorders (EDs) are psychiatric conditions characterized by a loss of control over food intake. The prevalence of anorexia nervosa (AN) is estimated at approximately 1-2%, while bulimia nervosa (BN) affects 2-3% of the population. EDs significantly impair functioning, have serious health consequences, and are associated with high mortality rates. Around 20% of patients with AN and 10% of those with BN develop a long-lasting illness, often referred to as Severe and Enduring Eating Disorders (SEED). While there is no scientific consensus on the definition of SEED, it is frequently defined as a duration of illness lasting seven years or more. Research suggests that factors maintaining EDs may differ from those that trigger them.

The underlying causes of EDs remain largely unknown, though their origins are considered multifactorial. Psychiatric comorbidities are highly prevalent in EDs, significantly influencing their course and outcomes. Personality disorders (PDs) are associated with poorer treatment outcomes for EDs, but longitudinal studies examining the trajectory of PDs in EDs are limited, and findings are inconsistent.

Dysfunctional emotion regulation (ER) has been identified as a transdiagnostic psychological risk factor for many psychiatric disorders, including EDs. ER difficulties can manifest as undercontrol, characterized by personality traits such as impulsivity and insufficient self-control, or overcontrol, characterized by emotional inhibition and excessive self-control och cognitive inflexibility. Some models propose that undercontrol is central to BN, while overcontrol are core features of AN. However, the course and stability of ER in EDs remain poorly understood due to a lack of longitudinal studies.

Another understudied factor in EDs is loneliness, encompassing perceived social isolation and a lack of connectedness. Loneliness has been linked to ER strategies, such as excessive self-control and emotional avoidance, which in youth can contribute to social isolation, reduced life satisfaction, and a higher risk of enduring mental health problems. The role of loneliness in SEED, however, is not well understood.

Further, research on EDs has proposed that biological factors, including dysregulation of the immune system, plays a role in the development and maintenance of the EDs. Studies indicate a pro-inflammatory state in AN, though it remains unclear whether this is a state or trait marker. The role of inflammation in BN is even less understood, and studies present mixed findings. Some evidence suggests an increased risk of BN in individuals with autoimmune or inflammatory diseases, highlighting the need for further investigation into inflammatory markers over the course of the illness.

In summary, clinical factors such as psychiatric comorbidity and personality disorders; psychological factors including personality characteristics, dysfunctional emotion regulation, overcontrol/undercontrol, cognitive inflexibility, loneliness, and severe eating disorder (ED) symptoms; and biological factors such as immune system dysregulation may all play a role in the development, maintenance, and relapse of EDs. However, research in this field is scarce.

This projects aims is to increase our knowledge about risk factors for a severe course in EDs. Our overarching research question is: What are the key clinical, psychological, and biological risk factors of a severe and enduring course of an eating disorder?

It is hypothesized that a chronic course of ED is related to severe ED symptoms, personality traits related to maladaptive over- and undercontrol, difficulties with emotion regulation (ER), and increased systemic inflammation.

Primary outcomes are

* eating disorder diagnosis at follow-up
* severity of eating disorder symptoms

Secondary outcomes are

* psychosocial impairment
* quality of life
* loneliness at follow-up
* comorbidity at follow-up
* systemic inflammatory activity at follow-up
* Physical status at follow-up

Predictors, moderators and mediators

* emotion regulation
* personality
* cognitive flexibility
* loneliness at baseline
* comorbidity at baseline
* systemic inflammatory activity at baseline
* duration of illness
* time in treatment
* motivation for change
* treatment completion/treatment dropout
* Physical status at baseline

PROCEDURE

Two prospective cohorts of patients with eating disorders (EDs)-one adolescent and one adult-will be followed longitudinally to examine changes in and the impact of clinical factors, personality traits, emotion regulation (ER) difficulties, loneliness, and biomarkers. Data will be collected at baseline, post-treatment, two years post-baseline, and at five, 10, and 20 years. Participants will be recruited consecutively from autumn 2024 onwards from the Eating Disorder Unit at the Uppsala Department of Child and Adolescent Psychiatry (ED-CAP) and the eating disorder unit for adults (ED-P).

Child and adolescent psychiatry (ED-CAP)

The eating disorder unit at the Department of Child and Adolescent Psychiatry at Uppsala University Hospital (CAP) treats patients with AN, BN, Other Specified Feeding or Eating Disorder (OSFED), and Avoidant Restrictive Food Intake Disorder (ARFID) up to 18 years. Patients are referred to the unit either by other healthcare professionals or by themselves and/or their parents.

All patients are systematically assessed using a structure implemented by Swedish ED clinics that provides valid data to the national quality register. The structure consists of an assessment of clinical history, diagnostic evaluation with the child and adolescent version of the MINI International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) or Electronic Psychiatric Screening Interview for children (EPSI-C), the Eating Disorder Examination interview (EDE-I), and clinician rating of symptoms and functioning (C-GAS) and the Clinical Global Impressions scale (CGI). In addition, weight and height are measured, and self-ratings with the Eating Disorder Examination Questionnaire (EDE-Q), Clinical Impairment Assessment Questionnaire (CIA), and Montgomery-Åsberg Depression Rating Scale Self-Assessment (MADRS-S) are collected.

After this initial assessment, all patients will be invited to participate in research. A research nurse will invite all patients and perform the initial somatic examination as well as sampling of blood. The patients who accept participation will sign informed consent to be included in the study. Since the youths are at least 14 years old, their parents/caregivers will also be required to accept participation and sign informed consent. Participants will receive questionnaires sent to them digitally.

The eating disorder clinic for adults (ED-P)

The eating disorder clinic for adults at the Department of Psychiatry at Uppsala University Hospital (ED-P) treats adults (≥ 18 years) with EDs. The clinic receives referrals from healthcare professionals (mainly physicians or psychologists) from other parts of the regional healthcare system. Patients can also refer themselves.

All patients undergo a systematic evaluation upon arrival at the eating disorder clinic. This consists of a clinical history and a structured diagnostic interview; either the MINI for DSM-5 or the Structured Clinical Interview for DSM-5 Axis I Disorders - Clinical Version (SCID-I CV). Patients also undergo the Eating Disorder Examination interview (EDE-I) and complete the self-report instruments Eating Disorder Examination Questionnaire (EDE-Q), Clinical Impairment Assessment Questionnaire (CIA), and Montgomery-Åsberg Depression Rating Scale Self-assessment (MADRS-S). Weight and height are measured.

All diagnostic assessments at the Department of Psychiatry are conducted by psychologists or physicians who have received training in the procedure. Patients who, during the assessment, are diagnosed with AN, BN, BED, ARFID, or OSFED of moderate to severe intensity, or OSFED with psychiatric comorbidity, and who accept treatment are accepted for treatment at P-ED. Patients who are diagnosed with mild OSFED or moderate OSFED without psychiatric comorbidity are referred to primary care for monitoring or treatment.

After this initial assessment, all patients will be invited to participate in research. An appointed person will invite all patients. If the patient accepts participation, they will sign an informed consent form. Participants will receive questionnaires sent to them digitally.

All Ages: Both ED-CAP and ED-P Participants will be asked about the collection of biomarkers through Uppsala Psychiatric Patient samples (UPP) (ethics approval Dnr 2012/081), which is an infrastructure for the collection of biological materials at the Department of Psychiatry at Uppsala University Hospital. All patients will be invited to participate in UPP, and inflammatory markers will be analyzed in accordance with the informed consent for UPP. Inflammatory markers will be analyzed from venous blood samples drawn from participants before treatment, immediately after treatment or dropout, and at the two-year follow-up.

At baseline, the following data will be collected: Diagnoses, physical examination (BMI, pulse, blood pressure), demographic characteristics, clinical characteristics, personality traits, psychological risk factors (e.g., ER difficulties, including loneliness), and biomarkers (including markers of inflammation). The same procedure will be repeated again after two years. A few questionnaires will be distributed at treatment termination or dropout.

After five, 10, and 20 years, patients will be followed up through National Helath registers and with questionnaires. Weighing will be performed weekly during treatment and at the follow-up two years later. At all time points, questionnaires will be distributed digitally. Process measures, such as the type of received treatment, number of treatment sessions, whether the patient dropped out or completed treatment, will be monitored. At follow-up, participants will be asked to answer a set of questions regarding, for example, living conditions, in addition to the questionnaires assessed at baseline.

QUALITY ASSURANCE PLAN

Interviewers will be trained and quality assured by calculating inter-rater agreement. For self-assessment, well established psychometrically evaluated instruments have been chosen. Special consideration has been given to selecting instruments suitable for both adolescents and adults.

SAMPLE SIZE ASSESSMENT

Sample size calculations were performed to ensure adequate power for the proposed analyses. With a Cohens effect size of d = 0.2, 199 participants will be required in each group, given an alpha of 0.05 and a power of 0.8. Dropout over time is expected, which increases as more time passes, estimating a 50% dropout by the final physical follow-up. Therefore, just under 400 participants need to be included in each group in order to have sufficient data for the last follow-up.

DATA ANALYSES

A range of statistical techniques will be employed to address the hypotheses and research aims, considering the longitudinal design, comparisons between the adolescent and adult cohorts, and diversity of outcome variables:

Descriptive analyses - Descriptive statistics (means, standard deviations, proportions) will summarize demographic, clinical, psychological, and biological variables at baseline and follow-up. Correlation analyses will explore relationships between predictors and primary and secondary outcomes.

Comparisons between subgroups

* Cluster analyses will be performed to identify subgroups of participants with different profiles of personality traits. These cluster will be compared regarding predictors, mediators/moderators, secondary outcomes, and primary outcomes.
* Between-group comparisons will also be conducted using t-tests, ANOVA or nonparametric alternatives (e.g., Mann-Whitney U tests) with regard to predictors and outcomes.

Longitudinal Regression Analyses

* Linear Mixed-Effects Models (LMM): These will evaluate changes in continuous outcomes over time.
* Generalized Estimating Equations (GEE): These models will analyze categorical outcomes, accounting for repeated measures and within-subject correlations.
* Logistic Regression: Logistic models will predict binary outcomes at follow-up.

Mediation and Moderation Analyses

* Mediation Analysis: mediation models will assess how variables mediate the relationship between predictors and primary and secondary outcomes.
* Moderation Analysis: Moderation models will explore how variables influence the relationship between predictors and primary and secondary outcomes.

Survival Analysis

- Cox proportional hazards models will be used to analyze time-to-event data, such as time to dropout and relapse.

Inflammatory Biomarker Analyses

- Levels of inflammatory markers in the ED samples will be compared to samples from individuals with other psychiatric disorders, as well as with healthy controls. Since blood samples will be taken upon repeated times during the study period, comparison of levels of inflammatory markers during disease course will be possible.

Missing data will be addressed as instructed for each instrument, ur by using multiple imputation or mixed-model approaches.

Subgroup Analyses

- Separate analyses will be conducted for adolescent and adult cohorts to examine potential differences in predictors and outcomes.

All statistical analyses will be performed using appropriate software (R, SPSS), and sensitivity analyses will be conducted to assess the robustness of findings.

ELIGIBILITY:
Inclusion criteria:

* found to meet the criteria for an eating disorder
* being in need of treatment
* having provided written informed consent (for minors, this includes consent from all caregivers and the minors themselves).

Exclusion criteria:

* Eating disorders symptoms in need of emergency care
* High risk for suicide
* An inability to respond to the questionnaires due to e.g., lack of knowledge in Swedish.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Two prospective cohorts of patients with ED, one adolescent and one adult, will be followed in terms of change in and impact of clinical factors, personality style, ER difficulties, loneliness, and biomarkers from baseline, after treatment, two years after baseline, and after five, 10 and 20 years. These cohorts will be consecutively recruited from 2024 onwards from the Eating Disorder Unit at the Uppsala Department of Child and Adolescent Psychiatry (CAP), from 14 to17 years of age, and the Uppsala Department of Psychiatry (P), from 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2048-12 (Estimated)

PRIMARY OUTCOMES:
Eating disorder examination interview (EDE-I) | At baseline and at two-year follow up
  EDE-I is a semi-structured interview for assessing symptoms of and diagnosing eating disorders, including providing information for grading severity according to e.g., the DSM 5. The EDE-I assesses a variety of eating disorder behaviors, weight control behaviors, and behavioral and cognitive features of eating disorder psychopathology.
Eating disorder Examination Questionnaire (EDE-Q) | At baseline, follow-up after treatment, and at 2, 5, 10, and 20 years follow-up.
  EDE-Q is a 28-item self-report questionnaire, designed to assess the range, frequency and severity of behaviors associated with an eating disorder. It is categorized into four sub-scales: Restraint, Eating Concern, Shape Concern and Weight Concern, and an overall global score. The score is obtained by calculating the mean for the total score and the subscales respectively (min = 0, max =6), higher scores indicate more severe eating disorder symptoms.
Eating Disorder-15 (ED-15) and for parents/caregivers (ED-15-P) | ED-15 at baseline, follow-up after treatment, and at 2, 5, 10, and 20 years follow-up (youth cohort only). ED-15-P At baseline, follow-up after treatment, and at 2 years follow-up.
  ED-15 assesses eating disorder attitudes and behaviors on a 15-item Likert scale, which includes 10 attitudinal items (scored from 0-6) and 5 items for frequency grading. ED-15-P include the same items but is answered by the youths caregiver instead. The ED-15 includes two attitudinal subscales: Weight & shape concerns and Eating concerns. The Overall attitudinal score is the mean of the scores on all ten items. Higher scores indicate more severe eating disorder symptoms.
Clinical Global Impression-Severity (CGI-S) | At baseline and at 2 year follow-up (youth cohort only).
  Global clinical rating of symptom severity on an 8-grade Likert scale (scored between 0-7). The CGI offers a clinician-determined summary that incorporates all available information, including the patient's history, psychosocial context, symptoms, behavior, and the impact of these symptoms on their functional ability. A higher score indicates a more severe psychopathology.
Eating disorder diagnosis during follow-up in registers | Registry data is retrieved at follow-up 5, 10 and 20 years
  Eating disorder diagnosis (AN, BN, BED, EDNOS, OSFED, UFED), collected from the National registries held by the National Board of Health and Welfare.

SECONDARY OUTCOMES:
Clinical Impairment Assessment questionnaire (CIA) | At baseline, follow-up after treatment, and at 2, 5, 10, and 20 years follow-up.
  The CIA is a 16-item self-report measure of the severity of psychosocial impairment due to eating disorder features, Each item is rated on a four-point Likert scale ranging from 'Not at all' to 'A lot'. The minimun score is zero and the maximum score is 48, with higher scores indicating a more severe impairment.
WHO Disability Assessment Schedule (WHODAS 2.0) | At baseline, follow-up after treatment, and at 2, 5, 10, and 20 years follow-up (adult cohort only).
  WHODAS 2.0 measure individual dysfunction in six domains of daily activities (cognition, mobility, self-care, relationships with people, life activities, and participation). It is measured on a five-point Likert scale ranging from no difficulty, to extreme difficulty. The score is calculated by dividing the total score with the number of items, resulting in a minimum score of zero and maximum score of 4. Higher scores indicate higher disability.
Uppsala scale of Functional Impairment in Daily life (UFID and UFID-P for parents) | UFID: At baseline, follow-up after treatment, and at 2, 5, 10, and 20 years follow-up (youth cohort only). UFID-P: At baseline, follow-up after treatment, and at 2 year follow-up.
  The UFID is a Five-item, five-point Likert scale that measures functional impairment in daily life on a score between 1-5. UFID-P includes the same items but is answered by the caregiver instead. Higher scores indicate more functional impairment.
Children's Global Assessment Scale (CGAS) | At baseline and at 2 year follow-up (youth cohort only).
  CGAS is a rating of general functioning for children and young people aged 4-16 years old. The clinician assesses a range of aspects of psychological and social functioning and gives the child or young person a single score between 1 and 100, based on their lowest level of functioning.
EQ-Visual Analogue Scale (EQ-VAS) | At baseline, follow-up after treatment, and at 2, 5, 10, and 20 years follow-up.
  The EQ-VAS is a vertical visual analogue scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health.
Social safeness and pleasure scale (SSPS) | At baseline, follow-up after treatment, and at 2, 5, 10, and 20 years follow-up.
  The SSPS is an 11-item self-rating instrument that assesses the extent to which people experience their world as safe, warm, and soothing, and how connected they feel to others. Participants indicate their answers on a five-point Likert scale, ranging from 1 (almost never) to 5 (almost all the time). Scores are added together to produce a total score in the range of 11-55, with higher scores representing higher perceived social safeness and connectedness to others.
  SSPS at baseline is a predictor/mediator/moderator, SSPS at follow-up is a secondary outcome.
Loneliness scale | At baseline, follow-up after treatment, and at 2, 5, 10, and 20 years follow-up.
  The Loneliness scale is an 11-item self-rating instrument includes a 6-item emotional subscale and a 5-item social subscale. Respondents are presented with a series of statements and asked to indicate the extent to which the statement applies to their situation on a four-point Likert scale. The total score can range between 0-11 with higher scores indicating greater feelings of loneliness.
  The Loneliness scale at baseline is a predictor/mediator/moderator, The Loneliness scale at follow-up is a secondary outcome.
UCLA Loneliness Scale | At baseline, follow-up after treatment, and at 2, 5, 10, and 20 years follow-up.
  UCLA Loneliness scale is a self-rating scale designed to measure ones subjective feelings of loneliness as well as feelings of social isolation. The scale comprises three questions that measure three dimensions of loneliness: relational connectedness, social connectedness and self-perceived isolation. Participants indicate their answers on a four-point Likert scale, providing a total score between 4-16, with higher scores indicating greater feelings of loneliness.
  The UCLA at baseline is a predictor/mediator/moderator, The UCLA at follow-up is a secondary outcome.
Montgomery Åsberg Depression Scale Self-assessment (MADRS-S) | At baseline, follow-up after treatment, and at 2, 5, 10, and 20 years follow-up.
  MADRS-S is a 9-item widely used self-rating measure of depressive severity. The intention of the scale is to give an image of the patients current state of mind. The patient grades how he/she felt during the last three days. Items are rated on a seven-point Likert scale, providing a total score between 0-54, with higher scores reflecting greater depression severity.
  The MADRS-S at baseline is a predictor/mediator/moderator, The MADRS-S at follow-up is a secondary outcome.
Comorbidity | At baseline, after treatment, and at 2 year follow-up (from medical journals) and at 10 and 20 years follow-up (from national health registers)..
  Comorbidity (including e.g., mood disorders, anxiety disorders, substance use disorders, and psychotic disorders) will be assess from medical journals, where diagnoses are based om the semi-structured interviews Electronic Psychiatric Screening Interview for children (EPSI-C), The Mini-International Neuropsychiatric Interview (M.I.N.I) for DSM-5 or the Structured Clinical Interview for DSM-5 Axis I Disorders - Clinical Version (SCID-I CV). Comorbidity will also be assessed from national health registers.
  Comorbidity at baseline is a predictor/mediator/moderator, comorbidity at follow-up is a secondary outcome.
Descriptive information about psychosocial functioning | Self-rated at baseline and at 2, 5, 10, and 20 years follow-up. Registry data is retrieved at follow-up 5, 10 and 20 years
  Occupation status
Descriptive information about psychosocial functioning | Self-rated at baseline and at 2, 5, 10, and 20 years follow-up. Registry data is retrieved at follow-up 5, 10 and 20 years
  Level of education
Descriptive information about psychosocial functioning | Self-rated at baseline and at 2, 5, 10, and 20 years follow-up. Registry data is retrieved at follow-up 5, 10 and 20 years
  Sick-leave
Descriptive information about psychosocial functioning | Self-rated at baseline and at 2, 5, 10, and 20 years follow-up. Registry data is retrieved at follow-up 5, 10 and 20 years
  Civil-status
Descriptive information about psychosocial functioning | Registry data is retrieved at follow-up 5, 10 and 20 years
  Number of children
Physical status - BMI | At baseline, weekly during treatment, follow-up after treatment, and at 2 year follow-up. Self-rated att 5, 10, and 20 year follow-up.
  Weight and height will be combined to report BMI in kg/m^2, assessed with a valid and reliable device in a standardized procedure.
  BMI at baseline is a predictor/mediator/moderator, BMI at follow-up is a secondary outcome.
Physical status - pulse | At baseline, and at 2 year follow-up.
  The number of times the heart beats within a certain time period. Pulse at baseline is a predictor/mediator/moderator, Pulse at follow-up is a secondary outcome.
Physical status - blood pressure | At baseline, and at 2 year follow-up.
  Blood pressure at baseline is a predictor/mediator/moderator, blood pressure at follow-up is a secondary outcome.

OTHER OUTCOMES:
The Avoidance and Fusion Questionnaire for Youth (AFQ-Y) | At baseline, follow-up after treatment, and at 2, 5, 10, and 20 years follow-up.
  The AFQ-Y is a self-rating instrument that measures psychological inflexibility. Participants rate their level of agreement on eight items on a 5-point Likert measuring one single factor. Score range is 0-24 and higher scores indicate a higher level of psychological inflexibility.
Emotion Regulation Questionnaire (ERQ) | At baseline, follow-up after treatment, and at 2, 5, 10, and 20 years follow-up.
  The ERQ is a self-rating instrument designed to assess individual differences in the use of emotion regulation strategies. It is composed of ten items divided into two factors: cognitive reappraisal and expressive suppression. Participants indicate their answers on a 7-point Likert-scale ranging from 1 (total disagreement) to 7 (total agreement).
Swedish universities Scale of Personality (SSP) | At baseline and at 2, 5, 10, and 20 years follow-up (adult cohort only).
  SSP is a self-report instrument assessing personality traits corresponding to biological correlates. It contains 91 items divided into 13 subscales. The scale can also be divided into a three-factor solution with Factor 1 reflecting Neuroticism; Factor 2 reflecting Aggressiveness; and Factor 3 reflecting Extraversion. Each item is given as a statement with a four-point response format, ranging from does not apply at all to applies completely. It is presented in standardized t-score ranging from 0-100 (mean 50 and standard deviation 10). Higher scorer indicate more pronounced characteristics of that specific trait.
Neuroticism-Extraversion-Openness Personality Inventory (NEO-PI) | At baseline, and at 2, 5, 10, and 20 years follow-up (youth cohort only)
  The NEO-PI is a self-report instrument designed to assess personality traits based on the Five-Factor Model of personality. It consists of 240 items grouped into five main domains: Neuroticism, Extraversion, Openness to Experience, Agreeableness, and Conscientiousness. Each domain is further divided into six specific facets, providing a detailed profile of personality traits. Responses are rated on a five-point Likert scale, ranging from "Strongly Disagree" to "Strongly Agree." Scores are typically presented as standardized T-scores, with higher scores indicating a stronger expression of the respective traits.
Ego Undercontrol Scale-13 (EUC-13) | At baseline and at 2, 5, 10, and 20 years follow-up
  EUC-13 is a 13 item self-rating instrument designed to assess personality types based on how people inhibit or express their emotional impulses, identifying over- and undercontrolled personality styles. It is answered on a four-point Likert-scale ranging from Disagree very strongly to Agree very strongly. The total score can range between 1-4, with higher scores indicating higher undercontrol and lower scores indicating higher overcontrol.
Ghrelin | At baseline and at 2 year follow-up
  Ghrelin will be analysed from blood samples. A solid phase sandwich enzyme linked immunosorbent assay (ELISA) (Mercodia AB, Uppsala, Sweden) will be used for the analyses.
Leptin | At baseline and at 2 year follow-up
  Leptin will be analysed from blood samples. A solid phase sandwich enzyme linked immunosorbent assay (ELISA) (Mercodia AB, Uppsala, Sweden) will be used for the analyses
Adinopectin | At baseline and at 2 year follow-up
  Adinopectin will be analysed from blood samples. A solid phase sandwich enzyme linked immunosorbent assay (ELISA) (Mercodia AB, Uppsala, Sweden) will be used for the analyses.
Inflammatory markers | At baseline and at 2 year follow-up
  Inflammatory markers will be analysed from blood samples. A panel of 100 different markers, will be anlyzed using an electrochemilumine-scence sandwich immunoassay, Meso Scale Discovery (K15049D and K15198D, Rockville, MD, USA) a multiplex platform.
Duration of illness | Duration of illness will be assessed via baseline data where the participant reports how old he/she was when the eating disorder began (baseline), as well as time passed from baseline (follow-up).
  How long the participant has had the eating disorder.
Time in treatment | This information will be gathered from self-reports (previous treatments) and patient journals (current treatment).
  Time spent in eating disorder treatment
Care utilization | Registry data is retrieved at follow-up 5, 10 and 20 years
  Days in hospital since baseline
Care utilization | Registry data is retrieved at follow-up 5, 10 and 20 years
  Received somatic and psychiatric care
Treatment completion/treatment droput | After treatment
  Data from medical journals will be reviewed to determine whether the treatment was completed as planned, prematurely terminated by the clinician's decision, or discontinued by the patient's decision.
Motivation for change | At baseline
  Participants are instructed to describe their goals for the eating disorder treatment they have sought. This description will be analyzed categorized in terms of motivation and compared to treatment outcomes and including completion or dropout from treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
Data will not be made publicly available due to confidentiality, but can be made available upon reasonable request to the corresponding author.

REFERENCES:
- [Background] Isaksson M, Ghaderi A, Wolf-Arehult M, Ramklint M. Overcontrolled, undercontrolled, and resilient personality styles among patients with eating disorders. J Eat Disord. 2021 Apr 16;9(1):47. doi: 10.1186/s40337-021-00400-0. PMID 33863394
- [Background] Gibson D, Mehler PS. Anorexia Nervosa and the Immune System-A Narrative Review. J Clin Med. 2019 Nov 8;8(11):1915. doi: 10.3390/jcm8111915. PMID 31717370
- [Background] Solmi M, Veronese N, Favaro A, Santonastaso P, Manzato E, Sergi G, Correll CU. Inflammatory cytokines and anorexia nervosa: A meta-analysis of cross-sectional and longitudinal studies. Psychoneuroendocrinology. 2015 Jan;51:237-52. doi: 10.1016/j.psyneuen.2014.09.031. Epub 2014 Oct 8. PMID 25462897
- [Background] Santini ZI, Pisinger VSC, Nielsen L, Madsen KR, Nelausen MK, Koyanagi A, Koushede V, Roffey S, Thygesen LC, Meilstrup C. Social Disconnectedness, Loneliness, and Mental Health Among Adolescents in Danish High Schools: A Nationwide Cross-Sectional Study. Front Behav Neurosci. 2021 Apr 12;15:632906. doi: 10.3389/fnbeh.2021.632906. eCollection 2021. PMID 33927599
- [Background] Hempel R, Vanderbleek E, Lynch TR. Radically open DBT: Targeting emotional loneliness in Anorexia Nervosa. Eat Disord. 2018 Jan-Feb;26(1):92-104. doi: 10.1080/10640266.2018.1418268. PMID 29384459
- [Background] Oldershaw A, Lavender T, Sallis H, Stahl D, Schmidt U. Emotion generation and regulation in anorexia nervosa: a systematic review and meta-analysis of self-report data. Clin Psychol Rev. 2015 Jul;39:83-95. doi: 10.1016/j.cpr.2015.04.005. Epub 2015 May 2. PMID 26043394
- [Background] Prefit AB, Candea DM, Szentagotai-Tatar A. Emotion regulation across eating pathology: A meta-analysis. Appetite. 2019 Dec 1;143:104438. doi: 10.1016/j.appet.2019.104438. Epub 2019 Aug 31. PMID 31479694
- [Background] Martinussen M, Friborg O, Schmierer P, Kaiser S, Overgard KT, Neunhoeffer AL, Martinsen EW, Rosenvinge JH. The comorbidity of personality disorders in eating disorders: a meta-analysis. Eat Weight Disord. 2017 Jun;22(2):201-209. doi: 10.1007/s40519-016-0345-x. Epub 2016 Dec 19. PMID 27995489
- [Background] Wentz E, Gillberg IC, Anckarsater H, Gillberg C, Rastam M. Adolescent-onset anorexia nervosa: 18-year outcome. Br J Psychiatry. 2009 Feb;194(2):168-74. doi: 10.1192/bjp.bp.107.048686. PMID 19182181
- [Background] Culbert KM, Racine SE, Klump KL. Research Review: What we have learned about the causes of eating disorders - a synthesis of sociocultural, psychological, and biological research. J Child Psychol Psychiatry. 2015 Nov;56(11):1141-64. doi: 10.1111/jcpp.12441. Epub 2015 Jun 19. PMID 26095891
- [Background] Keel PK, Brown TA. Update on course and outcome in eating disorders. Int J Eat Disord. 2010 Apr;43(3):195-204. doi: 10.1002/eat.20810. PMID 20186717
- [Background] Keski-Rahkonen A, Mustelin L. Epidemiology of eating disorders in Europe: prevalence, incidence, comorbidity, course, consequences, and risk factors. Curr Opin Psychiatry. 2016 Nov;29(6):340-5. doi: 10.1097/YCO.0000000000000278. PMID 27662598
- [Background] Treasure J, Duarte TA, Schmidt U. Eating disorders. Lancet. 2020 Mar 14;395(10227):899-911. doi: 10.1016/S0140-6736(20)30059-3. PMID 32171414